CLINICAL TRIAL: NCT04603664
Title: Role of Neutrophil Gelatinase-Associated Lipocalin (NGAL) and Cystatin C in Prediction of Acute Kidney Injury in Patients With Covid-19 Infection
Brief Title: Role of NGAL and Cystatin C in Prediction of Acute Kidney Injury Covid-19 Infection
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sanaa Farag Mahmoud Wasfy, lecturer of aneathesia, Ain Shams University
Other Study IDs: FMASU P82b/2020
Record Dates: First submitted 2020-10-17; First posted 2020-10-27 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Biochemical Markers ,NGAL,Cystatin c, Acute Kidneyinjury, Covid 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum refrigerated and divideded into 3 allicots for measurment of NGAL,cystatin c and creatinine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: blood sampling and measduring of serum NGAL and cystatin c on admission and after 48 hours and creatinine every day
  Interventions: Diagnostic Test: serum NGAL and cystatin c

INTERVENTIONS:
Diagnostic Test: serum NGAL and cystatin c — measuring serum NGAL and cystatin c on admission and after 48 hours in critically ill patients with covid 19 then compare results to serum creatinine and signs of acute kidney injury

SUMMARY:
Recent different biomarkers of acute kidney injury (AKI) have been manufactured by pharmaceutical industry. Studies proved that Neutrophil gelatinase-associated lipocalin (NGAL) and cystatin c are effective predictive biomarkers for early acute kidney injury in septic patients and in children after cardiopulmonary bypass. This study hypothesize that both cystatin c and Neutrophil gelatinase-associated lipocalin can predict AKI in patients with COVID-19 before elevation of serum urea and creatinine which may help early interference.

DETAILED DESCRIPTION:
Since December 2019, a novel coronavirus called SARSCoV-2 (severe acute respiratory syndrome coronavirus 2) has caused an international outbreak of respiratory illness described as COVID-19. Among 85 patients with COVID-19 an incidence of acute kidney injury was reported to be 23%. The kidney histology from autopsies of six patients showed severe acute tubular necrosis with macrophage and lymphocyte infiltration. Another important paper revealed prominent acute proximal tubular injury, accumulation of peritubular erythrocyte and glomerular fibrin microthrombi after autopsy. However, this kidney injury was not detected by routine measures (creatinine and/or BUN) in some patients denoting subclinical kidney injury. The pathophysiology of AKI associated with COVID-19 could be due to specific mechanisms such as direct cell injury from viral entrance through highly expressed renal ACE2 receptors. Also pro-inflammatory cytokines, an imbalanced renin-angotensin-aldosterone system and thrombotic events are accused in renal damage. Non-specific mechanisms include hypovolemia, haemodynamic changes, right heart failure, high levels of PEEP in mechanically ventilated patients, nephrotoxic drugs and nosocomial infections. A significant association between kidney failure and death was documented in five studies. Hypoxemia and impairment of gas exchange has been identified as elements associated with AKI in patients with acute respiratory distress syndrome (ARDS).

Studies focusing on AKI with COVID-19 are needed urgently in order to identify the mechanism of renal affection and to predict the risk of AKI. Pharmaceutical industries with academia have made a lot of progress in the field of sensitive and specific preclinical biomarkers of kidney injury. Neutrophil gelatinase-associated lipocalin (NGAL) is composed of 178 amino acids. this glycoprotein is reabsorbed in the proximal tubules after its filtration through the glomeruli.

In a mouse model of renal ischemia, NGAL gene was rapidly expressed and upregulated within 3 hours of injury. The NGAL mRNA level increased more than 1000-fold 24-48 hours after injury. Thus, NGAL can be a useful tool to diagnose infection mediated AKI. Nonglycosylated Cystatin C is a protein produced by nucleated cells at constant rate. It is easily filtered through the glomeruli due to its positive charge at physiological pH and its low molecular weight. Then, it is reabsorbed and completely catabolized in the proximal tubules. Use of serum cystatin C as a marker of glomerular filtration rate (GFR) is well documented, and some authors have suggested that it may be more accurate than serum creatinine for this purpose. Complete evaluation of the clinical and laboratory picture of COVID-19 associated AKI is crucial to design preventive strategies and to suggest targeted interventions

ELIGIBILITY:
Inclusion Criteria:

* person with the one of the following symptoms: fever and respiratory symptoms with radiological findings of pneumonia compatible with COVID-19

  1. Respiratory distress (≥ 30 breaths/ min);
  2. Oxygen saturation ≤ 93% at rest;
  3. Arterial partial pressure of oxygen (PaO2)/ fraction of inspired oxygen (FIO2) ≤ 300.
  4. Cases with chest imaging that shows obvious lesion progression within 24-48 hours > 50%.
  5. Respiratory failure and requiring mechanical ventilation;
  6. Shock;
  7. other organ failure that requires ICU care.

Exclusion Criteria:

* patients classified as mild corona virsus disease, patients with end-stage renal disease (ESRD) or on chronic regular dialysis, presence of AKI and anuria at the time of ICU admission, history of chronic kidney disease, severe urinary tract infection, kidney malignancy, and renal transplantation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients from 18-85 diagnosed as covid 19 infection by nasaopharyngeal swap
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
measure both cystatin c and Neutrophil gelatinase-associated lipocalin on admission and after 48 hours. (NGAL) as recent biomarkers in prediction of AKI in patients with COVID-19. | 12 days starting from hospital admission
  biochmical tests for detection of NGAL and Cystatin c in crirically ill Covid 19 patients

SECONDARY OUTCOMES:
development of acute kidney injury lipocalin (NGAL) to AKI severity and prognosis of AKI in patients with COVID-19 infection | 12 days starting from day of admission
  increased serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: sanaa wasfy, Principal Investigator — lecturer
Locations (2):
- Egypt (2):
  - Ainshams hospitals, Cairo
  - Sanaa Wasfy, New Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diao, C.H. Wang, R.S. Wang, Z.Q. Feng, Y.J. Tan, H.M. Wang, et al. ( 2020 ) Human kidney is a target for novel severe acute respiratory syndrome coronavirus 2[SARS-CoV-2] infection [preprint posted online April 10, . medRxiv doi:10.1101/2020.03.04.20031120 Xu S, Fu L, Fei J et al (2020) Acute kidney injury at early stage as a negative prognostic indicator of patients with COVID-19: a hospital-based retrospective analysis. medRxiv 2020.03.24.20042408. https://doi.org/10.1101/2020.03.24.20042408 Darmon M, Schortgen F, Leon R et al (2009) Impact of mild hypoxemia on renal function and renal resistive index during mechanical ventilation. Intensiv Care Med 35:1031-1038. https://doi.org/10.1007/s00134-008-1372-5 Darmon M, Schortgen F, Leon R et al (2009) Impact of mild hypoxemia on renal function and renal resistive index during mechanical ventilation. Intensiv Care Med 35:1031-1038. https://doi.org/10.1007/s00134-008-1372-5